CLINICAL TRIAL: NCT07229235
Title: REAL-CARE: Real-world Effectiveness of iptacopAn in itaLian Patients With Paroxysmal noCturnAl HemoglobinuRia: an Observational Study
Brief Title: REAL-CARE: Real-world Effectiveness of Iptacopan in Italian Patients With Paroxysmal Nocturnal Hemoglobinuria
Acronym: REAL-CARE
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023C1IT01
Record Dates: First submitted 2025-10-30; First posted 2025-11-14 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: REAL-CARE; ptacopan; paroxysmal nocturnal hemoglobinuria; PNH; NIS
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Iptacopan: Treatment with iptacopan

SUMMARY:
This study evaluates iptacopan effectiveness and safety in routine clinical practice, with a focus on hematological response, transfusion avoidance, and patient-reported outcomes.

The primary objective of the REAL-CARE study is to is to assess the long-term hematological response following iptacopan initiation. This will be assessed through the absolute change in hemoglobin (Hb) levels at 12 months post-initiation, and the proportion of patients who remain free from red blood cell (RBC) transfusions, prescribed as per local requirement and based on Investigator's judgment, from Day 14 through Month 12 after starting iptacopan.

DETAILED DESCRIPTION:
This is a local, multicenter, observational study with retrospective, retro-prospective and prospective cohorts. Adult patients with PNH either naïve to iptacopan or transitioning from the Managed Access Program (MAP) starting from January 2023 will be enrolled. Primary data will be collected prospectively; secondary data will be retrieved retrospectively from patients previously treated under MAP. A mix of primary and secondary data will be collected in retro-prospective patients. Patients will be indexed on the date of iptacopan initiation and will be followed up for 24 months or until iptacopan discontinuation (due to occurrence of an adverse event, lack of efficacy etc), clinical decision, death, administrative issues, consent withdrawal or loss to follow-up, whichever comes first. The enrollment period is planned to last 15 months, with potential adjustments based on enrollment progress. No treatment decision will be influenced by study participation.

No extra visits, examinations, or procedures are imposed. Questionnaires should be collected at the indicated timepoints whenever possible, but, since the administration of the questionnaires represents an additional procedure not included in routine clinical care, these timepoints are considered indicative only, and patients will not be recalled specifically to complete questionnaires if a routine clinical visit is not scheduled.

ELIGIBILITY:
Inclusion criteria:

1. signed informed consent: patient must provide written informed before any study assessment is collected; in case of deceased patients, informed consent is not required as per Art. 110, comma 1 of Legislative Decree n° 196, dated 30 June 2003 as amended by D.lgs. 101/2018 and the "Autorizzazione generale al trattamento dei dati personali effettuato per scopi di ricerca scientifica" n° 9/2016
2. Male and female,
3. ≥ 18 years of age,
4. documented diagnosis of PNH,
5. followed in Italian clinical sites,
6. on treatment with iptacopan prescribed as per routine medical care (i.e. patients naïve to treatment for whom the decision to start this treatment has already been made on the basis of clinical practice and according to SmPC and AIFA criteria and regardless of inclusion in this study or patients already treated under the Managed Access Program (MAP))

Exclusion criteria:

1.Concomitant participation in an interventional clinical study related to PNH or its treatment.

No other inclusion/exclusion criteria apply other than the requirements stated in the Summary of Product Characteristics (SmPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Italian population of adult patients with PNH either naïve to iptacopan or transitioning from the Managed Access Program (MAP) starting from January 2023
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
absolute change in Hb level post iptacopan initiation | 12 months
  12-month absolute change in hemoglobin (Hb) level post iptacopan initiation
Proportion of patients with no RBC transfusions | 12 months
  12-month proportion of patients with no Red Blood Cells (RBC) transfusions, prescribed as per local requirement and based on Investigator's judgment, after Day 14.

SECONDARY OUTCOMES:
Socio-demographic and clinical variables of Paroxysmal Nocturnal Hemoglobinuria population | date of iptacopan start, day 0
  Descriptive measures of the socio-demographic variables, proportion of PNH cells, clinical symptoms, laboratory parameters, concomitant diseases and treatments and outcomes of PNH patients at iptacopan initiation.
Absolute change in Hb level post iptacopan initiation | date of iptacopan start (day 0), 24 months
  24-month absolute change in Hb level post iptacopan initiation
Proportion of patients who didn't need RBC transfusion | 24 months
  24-month proportion of patients who didn't need RBC transfusion, prescribed as per local requirement and based on Investigator's judgment, post iptacopan initiation
Proportion of patients with Hb levels ≥ 12 g/dL AND no RBC transfusion | 12 month, 24 month
  12- and 24-month proportion of patients with Hb levels ≥ 12 g/dL AND no RBC transfusion, prescribed as per local requirement and based on Investigator's judgment, between Day 14 and month 12 or month 24
Proportion of patients with change in Hb levels ≥ 2 g/dL post iptacopan initiation AND no RBC transfusion | 12 month, 24 month
  12- and 24-month proportion of patients with change in Hb levels ≥ 2 g/dL post iptacopan initiation AND no RBC transfusion, prescribed as per local requirement and based on Investigator's judgment, between Day 14 and month 12 or month 24
Average number of RBC transfusion | 12 months and 24 months
  Average number of RBC transfusion, prescribed as per local requirement and based on Investigator's judgment, per patient during 12- and 24-months post iptacopan initiation
Percentage change in LDH level post iptacopan initiation | date of iptacopan start (day 0), month 12, month 24
  12- and 24-month percentage change in LDH level post iptacopan initiation.
Change in reticulocyte count post iptacopan initiation. | date of iptacopan start (day 0), month 12, month 24
  12- and 24-month change in reticulocyte count post iptacopan initiation.
Absolute change in bilirubin level post iptacopan initiation. | date of iptacopan start (day 0), month 12, month 24
  12- and 24-month absolute change in bilirubin level post iptacopan initiation.
Frequency of adverse events (AE) and serious adverse events (SAE) over 12 and 24 months of follow-up | 12 months and 24 months
  Frequency of adverse events (AE) and serious adverse events (SAE) over 12 and 24 months of follow-up post iptacopan initiation
Proportion of BTH occurrence | 12 months and 24 months
  Proportion of Breakthrough Hemolysis (BTH) occurrence over 12 and 24 months of follow-up post iptacopan initiation
Type and proportion of Infections occurrence over 12 and 24 months of follow-up | 12 months and 24 months
  Type and proportion (count and percentage) of Infections occurrence over 12 and 24 months of follow-up post iptacopan initiation
Type and proportion of major adverse vascular events (MAVEs) occurrence | 12 months and 24 months
  Type and proportion of major adverse vascular events (MAVEs) occurrence over 12 and 24 months of follow-up post iptacopan initiation
Type and proportion of new comorbidities | 12 months and 24 months
  Type and proportion of new comorbidities occurred within 12 and 24 months of follow-up post iptacopan initiation
Type and proportion of concomitant medications newly prescribed | 12 months and 24 months
  Type and proportion of concomitant medications newly prescribed during 12 and 24 months of follow-up post iptacopan initiation
Absolute change in Medication Adherence Report Scale - 5 item (MARS-5) scores | date of iptacopan start (day 0), month 12 and month 24
  The MARS-5 questionnaire is a validated self-report questionnaire developed to assess patient adherence to prescribed medication, focusing on both intentional and unintentional non-adherence.
  It consists of five items, each rated on a 5-point Likert Scale, from 0 ("Always") to 5 ("Never").
  Items evaluate behaviors such as forgetting to take medications, altering the dose or stopping the treatment. The total score ranges from 5 to 25, with higher scores indicating better adherence to treatment.
Absolute change from iptacopan initiation in PROMIS-29+2 score. | date of iptacopan start (day 0), month 12 and month 24
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Profile-29+2 is a validated standardized patient reported outcome measure to assess generic health-related quality of life. The questionnaire covers the following nine health domains: Physical function, Anxiety, Depression, Fatigue, Sleep disturbance, Ability to participate in social roles and activities, Pain interference, Cognitive function and Pain intensity.
  The recall period for all items is the past 7 days. Each of the first eight domains is assessed through 4 items using a 5-point Likert scale. Pain intensity is measured with a single item on an 11-point numeric rating scale from 0 ("no pain") to 10 ("worst imaginable pain").
  Each domain is scored separately, with T-scores used to represent the severity or level of functioning in each area. Higher scores can indicate either better health (e.g., physical function) or greater severity of symptoms (e.g., anxiety, depression).
Absolute change from iptacopan initiation in WPAI:SHP score. | date of iptacopan start (day 0), month 12 and month 24
  Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) is a validated patient-reported outcome measure designed to assess the impact of a specific health problem on work and daily activities. In this study, the questionnaire has been customized for PNH. It includes six questions grouped into four key domains: Absenteeism (work time missed due to PNH), Presenteeism (impairment while working due to PNH), Overall work productivity loss (combined absenteeism and presenteeism), Activity impairment (impact of PNH on regular daily activities outside of work).
  The recall period is the past 7 days. Responses are used to calculate the percentage of work time missed and the level of impairment experienced by the patient. Higher scores represent greater impairment and reduced productivity.
Number of hospitalizations, emergency room visits, and hospital-based outpatient visits attributable to the management of AEs related to the study treatment | Up to 24 months
  Healthcare resources utilization:
  The number of hospitalizations, emergency room visits, and hospital-based outpatient visits attributable to the management of adverse events (AEs) related to the study treatment will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No